CLINICAL TRIAL: NCT00005514
Title: Dietary Patterns and Risk of Cardiovascular Disease
Status: Completed | Type: Observational
Sponsor: Harvard School of Public Health (HSPH) (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Frank B. Hu, Professor, Harvard School of Public Health (HSPH)
Other Study IDs: 5032; R01HL060712 (NIH)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2013-03-20 (Estimated); Status verified 2013-03

CONDITIONS: Cardiovascular Diseases; Coronary Disease; Cerebrovascular Disorders; Heart Diseases; Cerebrovascular Accident
MeSH Terms: conditions — Cardiovascular Diseases; Coronary Disease; Cerebrovascular Disorders; Heart Diseases; Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Plasma and buffy coat

SUMMARY:
To study, prospectively, the association between dietary patterns and risk of coronary heart disease (CHD), ischemic stroke, and hemorrhagic stroke in cohort studies of 121,700 women age 30 to 55 years at baseline in 1976 (the Nurses; Health Study; NHS) and 51,529 men aged 40-75 years at baseline in 1986 (the Health Professionals Follow-up Study; HPFS).

DETAILED DESCRIPTION:
DESIGN NARRATIVE:

In the first five years of the study analyses were performed on food consumption data collected through semiquantitative food frequency questionnaires at baseline and during follow-up in the Nurses Health Study and Health Professionals Follow-up Study cohorts. Dietary patterns were derived from the food consumption data using factor analysis, cluster analysis, and dietary indexes (based on prevailing dietary recommendations). In addition, using existing datasets from dietary validation studies in sub-samples of the two cohorts, the reproducibility and validity of dietary patterns defined by factor/cluster analysis and dietary indexes were evaluated. Further, using prospectively collected and stored bloods in the NHS (n-32,826) during 1989-1990 and the HPFS (n-18,000) during 1993-1994, the investigators examined whether observed associations between dietary patterns and CHD were explained by (or mediated through) plasma biochemical measurements (including serum lipids, thrombotic factors, antioxidants, fasting insulin, and homocysteine levels) in a nested case-control design; and they assessed prospectively the relationship between dietary patterns and these biomarkers in the control samples.

The study was renewed in 2005 to apply novel statistical methods (such as confirmatory factor analysis and structural equation modeling) to validate various dietary patterns and examine their associations with risk of type 2 diabetes, cardiovascular disease and total mortality in two large ongoing cohort studies, the Nurses' Health Study (n=121,700) and Health Professionals' Follow-up Study (n=51,529). In addition to evaluating prevailing dietary recommendations, the study will also examine the role of the Mediterranean-type dietary pattern, the Dietary Approaches to Stop Hypertension (DASH) dietary pattern, and the Atkins-type diet in predicting health outcomes. Using repeated measurements of diet, the study will examine the impact of changes in eating patterns and diet quality over time on subsequent risk of diabetes, CVD, and total mortality. In addition, it will examine relationships between major dietary patterns and novel plasma biomarkers of inflammation and endothelial function and whether such relationships are mediated through obesity. Finally, the study will test interactions between dietary patterns and individual single nucleotide polymorphisms (SNPs) and haplotypes of several promising candidate genes in the inflammation and endothelial dysfunction pathway on risk of coronary heart disease, including PPARa, PPARy, Adiponectin (AdipoQ), PON1, IL-6, TNF-a, ICAM-1, VCAM-1, E-Selectin, NOS3, ACE gene, and angiotensinogen (ANG) genes.

ELIGIBILITY:
no history of chronic diseases at baseline

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Nurses' Health Study and Health Professionals' Follow-up Study
Sampling Method: Non-Probability Sample
Enrollment: 120000 (Actual)
Dates: Start 1998-08; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
Incident cardiovascular disease | 1980-2008
  Myocardial infarction, fatal coronary disease, and stroke documented by medical records

REFERENCES:
- [Background] Hu FB, Rimm EB, Stampfer MJ, Ascherio A, Spiegelman D, Willett WC. Prospective study of major dietary patterns and risk of coronary heart disease in men. Am J Clin Nutr. 2000 Oct;72(4):912-21. doi: 10.1093/ajcn/72.4.912. PMID 11010931
- [Background] Hu FB, Stampfer MJ, Manson JE, Grodstein F, Colditz GA, Speizer FE, Willett WC. Trends in the incidence of coronary heart disease and changes in diet and lifestyle in women. N Engl J Med. 2000 Aug 24;343(8):530-7. doi: 10.1056/NEJM200008243430802. PMID 10954760
- [Background] Digranes A, Hardardottir H, Bottolfsen KL. Temafloxacin: in vitro comparison with five other antibacterial agents. Chemotherapy. 1991;37(2):98-105. doi: 10.1159/000238840. PMID 2032475
- [Background] Hu FB, Rimm E, Smith-Warner SA, Feskanich D, Stampfer MJ, Ascherio A, Sampson L, Willett WC. Reproducibility and validity of dietary patterns assessed with a food-frequency questionnaire. Am J Clin Nutr. 1999 Feb;69(2):243-9. doi: 10.1093/ajcn/69.2.243. PMID 9989687
- [Background] McCullough ML, Feskanich D, Stampfer MJ, Rosner BA, Hu FB, Hunter DJ, Variyam JN, Colditz GA, Willett WC. Adherence to the Dietary Guidelines for Americans and risk of major chronic disease in women. Am J Clin Nutr. 2000 Nov;72(5):1214-22. doi: 10.1093/ajcn/72.5.1214. PMID 11063452
- [Background] Fung TT, Rimm EB, Spiegelman D, Rifai N, Tofler GH, Willett WC, Hu FB. Association between dietary patterns and plasma biomarkers of obesity and cardiovascular disease risk. Am J Clin Nutr. 2001 Jan;73(1):61-7. doi: 10.1093/ajcn/73.1.61. PMID 11124751
- [Background] Fung TT, Willett WC, Stampfer MJ, Manson JE, Hu FB. Dietary patterns and the risk of coronary heart disease in women. Arch Intern Med. 2001 Aug 13-27;161(15):1857-62. doi: 10.1001/archinte.161.15.1857. PMID 11493127
- [Background] Hu FB, Willett WC. Optimal diets for prevention of coronary heart disease. JAMA. 2002 Nov 27;288(20):2569-78. doi: 10.1001/jama.288.20.2569. PMID 12444864
- [Background] Osganian SK, Stampfer MJ, Rimm E, Spiegelman D, Manson JE, Willett WC. Dietary carotenoids and risk of coronary artery disease in women. Am J Clin Nutr. 2003 Jun;77(6):1390-9. doi: 10.1093/ajcn/77.6.1390. PMID 12791615
- [Background] Hu FB. Plant-based foods and prevention of cardiovascular disease: an overview. Am J Clin Nutr. 2003 Sep;78(3 Suppl):544S-551S. doi: 10.1093/ajcn/78.3.544S. PMID 12936948
- [Background] Osganian SK, Stampfer MJ, Rimm E, Spiegelman D, Hu FB, Manson JE, Willett WC. Vitamin C and risk of coronary heart disease in women. J Am Coll Cardiol. 2003 Jul 16;42(2):246-52. doi: 10.1016/s0735-1097(03)00575-8. PMID 12875759
- [Background] Halton TL, Hu FB. The effects of high protein diets on thermogenesis, satiety and weight loss: a critical review. J Am Coll Nutr. 2004 Oct;23(5):373-85. doi: 10.1080/07315724.2004.10719381. PMID 15466943
- [Background] Fung TT, Stampfer MJ, Manson JE, Rexrode KM, Willett WC, Hu FB. Prospective study of major dietary patterns and stroke risk in women. Stroke. 2004 Sep;35(9):2014-9. doi: 10.1161/01.STR.0000135762.89154.92. Epub 2004 Jul 1. PMID 15232120
- [Background] Schulze MB, Hoffmann K, Manson JE, Willett WC, Meigs JB, Weikert C, Heidemann C, Colditz GA, Hu FB. Dietary pattern, inflammation, and incidence of type 2 diabetes in women. Am J Clin Nutr. 2005 Sep;82(3):675-84; quiz 714-5. doi: 10.1093/ajcn.82.3.675. PMID 16155283
- [Background] Hu FB. Protein, body weight, and cardiovascular health. Am J Clin Nutr. 2005 Jul;82(1 Suppl):242S-247S. doi: 10.1093/ajcn/82.1.242S. PMID 16002829